CLINICAL TRIAL: NCT02660229
Title: A 5-day, Multicentre, Randomized, Open-label, Parallel Group, Active Control Pilot Study to Evaluate the Efficacy and Safety of OxyNorm® (Oxycodone Hydrochloride Injection) in Comparison With Morphine Sulfate Through the IV Continuous Infusion Regimen in Patients With Cancer Pain
Brief Title: An Interventional Study for Patient With Cancer Pain to Evaluate the Efficacy and Safety of OxyNorm® Compared to Morphine Sulfate Through the IV Continuous Infusion.
Acronym: SWITCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OXI15-KR-401
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-04

CONDITIONS: Cancer Pain
Keywords: Intravenous injection in cancer pain
MeSH Terms: conditions — Cancer Pain | interventions — Oxycodone; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone Hydrochloride (Experimental): Brand Name: OxyNorm® Generic name: Oxycodone hydrochloride
  Interventions: Drug: Oxycodone Hydrochloride
- Morphine Sulphate (Active Comparator): Brand name: BC Morphine sulfate Generic name: Morphine sulfate
  Interventions: Drug: Morphine Sulphate

INTERVENTIONS:
Drug: Oxycodone Hydrochloride — Oxycodone injection
  Other Names: Oxynorm
  Arms: Oxycodone Hydrochloride
Drug: Morphine Sulphate — Morphine sulphate injection
  Other Names: BC morphine
  Arms: Morphine Sulphate

SUMMARY:
The purpose of this study is to compare of difference in NRS scores from baseline to the completion of treatment (5 days) in patients with administration of morphine sulfate versus oxycodone hydrochloride.

DETAILED DESCRIPTION:
5days, Multi-centers, Randomization, Open label, Parallel, Active Comparator, Phase 4 Study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women aged 19 years or more
2. Patients with cancerous pain who are hospitalized or scheduled for hospitalization at Screening and not planned to be discharged during the study
3. Patients with mean moderate to severe pain over the past 7 days at Screening as verbally confirmed (NRS 4 or higher)
4. Subjects who voluntarily signed the Informed Consent Form for the study
5. Subjects who are capable of understanding details of the study and verbal communication on pain intensity

Exclusion Criteria:

1. Patients who reached the narcotic analgesic dose corresponding to the followings for cancerous pain treatment immediately prior to Screening (oral morphine dose 195mg/day, oral oxycodone dose 130mg/day, patch fentanyl dose 75μg/hour)
2. Patients with a medical history of hypersensitivity to an ingredient of oxycodone hydrochloride or morphine sulfate or other narcotic analgesics
3. Patients who have contraindications and cautions when study drugs administered.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinhyong Kang, Dr. Ph.D, Principal Investigator — Seoul St. Mary's Hospital, The Catholic University of Korea
Locations (1):
- Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee KH, Kang JH, Oh HS, Choi MK, Shim BY, Eum YJ, Park HJ, Kang JH. Intravenous Oxycodone versus Intravenous Morphine in Cancer Pain: A Randomized, Open-Label, Parallel-Group, Active-Control Study. Pain Res Manag. 2017;2017:9741729. doi: 10.1155/2017/9741729. Epub 2017 Oct 31. PMID 29670416

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxycodone Hydrochloride: Brand Name: OxyNorm® Generic name: Oxycodone hydrochloride
  Oxycodone Hydrochloride: Oxycodone injection. The 10mg/1ml or 20mg/2ml was injected through intravenous PCA according to patient's pain intensity
- Morphine Sulphate: Brand name: BC Morphine sulfate Generic name: Morphine sulfate
  Morphine Sulphate: Morphine sulphate injection. The 5mg/5ml or 30mg/2ml was injected through intravenous PCA according to patient's pain intensity.
Period: Overall Study
Arm/Group | Oxycodone Hydrochloride | Morphine Sulphate
Started | 34 (Randomization) | 32 (Randomization)
Safety Analysis Set | 34 | 32
FAS Set | 33 (Oxycodone group: 1 patient was missed any efficacy assessment.) | 32
Per Protocol Set | 28 (Adverse events N=1, Prohibited medication N=4) | 29 (Withdrawal of ICF N=1, IC/EC deviation N=1, Prohibited medication N=1)
Completed | 32 | 31
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic data was analysed FAS set.
Groups:
- Oxycodone Hydrochloride: Brand Name: OxyNorm® Generic name: Oxycodone hydrochloride
  Oxycodone Hydrochloride: Oxycodone IV injection
- Morphine Sulphate: Brand name: BC Morphine sulfate Generic name: Morphine sulfate
  Morphine Sulphate: Morphine sulphate IV injection
- Total: Total of all reporting groups
Arm/Group | Oxycodone Hydrochloride | Morphine Sulphate | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Customized [Number; unit: participants]
  <39 years | 0 | 2 | 2
  40-49 years | 1 | 2 | 3
  50-59 years | 5 | 6 | 11
  60-69 years | 27 | 22 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 21 | 22 | 43
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change in the Mean Pain Score(NRS) From Baseline(Day 0) to Day 5.
Description: For the pain assessment value for efficacy assessment, Subjects perform pain grading through Numeric rating score(NRS) from 1 to 10 for the mean pain intensity over the past 7 days at Screening, and mean pain intensity over the past 24 hours at Baseline (Day 0), Day 1, Day 2, Day 3, Day 4, Day 5.
  Verbal measurement can be conducted by subjects without using visual data. '0' indicates 'no pain', and as the number increases, the pain gets more severe, and '10' indicates the worst pain.
Time Frame: 5 days
Population: Primary endpoint was analysed FAS set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxycodone Hydrochloride | Morphine Sulphate
Number analyzed (Participants) | 33 | 32
units on a scale | -3.52 (2.17) | -3.13 (1.84)

2. Secondary Outcome: Total Dose of IV(IV Infusion+Bolus Injection) Study Drug Administered During the Treatment Duration
Description: The dose of the study drugs intravenously administered was checked and recorded every day. The information on the dose administered from baseline to each assessment time point was collected based on records on the chart, and in the event of dose change/end of treatment, pertinent date and time, and dose were recorded accurately on the chart.
  ‡ Total administered dose of the study drugs (mg)= IV infusion (mg/hr) * [(End date - start date) * 24 + (end time - start time)] + bolus injection (mg)
Time Frame: 5 days
Population: FAS set.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Oxycodone Hydrochloride | Morphine Sulphate
Number analyzed (Participants) | 33 | 32
mg | 226.80 (110.44) | 226.64 (135.13)

3. Secondary Outcome: Patient's Overall Satisfaction With Each Continuous Infusion on Day 5 After Randomization
Description: The subjects made an assessment of overall treatment satisfaction regarding pain using the PGI-C on a 7-point scale (1: Very much improved, 2: Much improved, 3: Minimally improved, 4: No change, 5: Minimally worse, 6: Much worse, 7: Very much worse) after baseline and at the end of the study (Day 5).
Time Frame: 5 days
Population: FAS set. However, OxyNorm 1 subject (S08-09) and Morphine sulfate 1 subject (S08-15) were not assessed on Day 5 after baseline. So, missing data was excluded from analysis. Oxynorm group 32 subjects and Morphine group 31 subjects were analysed for PGIC.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxycodone Hydrochloride | Morphine Sulphate
Number analyzed (Participants) | 32 | 31
Participants
  1:Very much improved | 9 | 8
  2: Much Improved | 10 | 10
  3: Minimally improved | 12 | 12
  4: No change | 1 | 1
  5: Minimally worse | 0 | 0
  6: Much worse | 0 | 0
  7: Very much worse | 0 | 0

4. Secondary Outcome: Investigator's Overall Satisfaction With IV Infusion on 5 Days After Randomization
Description: The investigators made an assessment using the CGI-C on a 7-point scale (1: Very much improved, 2: Much improved, 3: Minimally improved, 4: No change, 5: Minimally worse, 6: Much worse, 7: Very much worse).
Time Frame: 5 days
Population: FAS set. However, OxyNorm 1 subject (S08-09) and Morphine sulfate 1 subject (S08-15) were not assessed on Day 5 after baseline.
  So, the data was missed.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxycodone Hydrochloride | Morphine Sulphate
Number analyzed (Participants) | 32 | 31
Participants
  1: Very much improved | 10 | 9
  2: Much improved | 16 | 15
  3: Minimal improved | 5 | 6
  4. No change | 1 | 1
  5. Minimally worse | 0 | 0
  6. Much worse | 0 | 0
  7. Very much worse | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 days
Description: The safety analysis was performed regarding AEs, vital signs, physical examination, clinical laboratory test, and ECG in the Safety set involving all subjects who received the study drug after randomization in this clinical study.
Arm/Group | Oxycodone Hydrochloride | Morphine Sulphate
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 3/34 | 2/32
Other Adverse Events (participants affected / at risk) | 14/34 | 11/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone Hydrochloride (N=34) | Morphine Sulphate (N=32)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone Hydrochloride (N=34) | Morphine Sulphate (N=32)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (5) — Adverse drug reaction
Constipation (Gastrointestinal disorders) | 7 (7) | 3 (3) — Adverse drug reaction
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Adverse drug reaction
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Adverse drug reaction
Asthenia (General disorders) | 0 (0) | 1 (1) — Adverse drug reaction
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) — Adverse drug reaction
Somnolence (Nervous system disorders) | 3 (3) | 1 (1) — Adverse drug reaction
Sedation (Nervous system disorders) | 1 (1) | 0 (0) — Adverse drug reaction
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Adverse drug reaction
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Adverse drug reaction
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) — Adverse drug reaction
Hypotension (Vascular disorders) | 1 (1) | 0 (0) — Adverse drug reaction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No